CLINICAL TRIAL: NCT05839522
Title: Australian Hepatitis and Risk Survey in Prisons
Acronym: AusHep
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kirby Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: VISP1901
Record Dates: First submitted 2023-03-06; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Hepatitis C; Hepatitis B; HIV Infections
Keywords: Blood-borne viruses; Prisons; Surveillance
MeSH Terms: conditions — Hepatitis C; Hepatitis B; HIV Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Persons in custody in Australia: Representative sample of 2400 people in prison from 25 representative prisons in Australia will participate in a biobehavioural survey involving point-of-care testing for HCV antibodies and RNA (if antibody positive), HBV surface antigens and antibodies, and HIV antibodies, and an interview-style survey.
  Interventions: Diagnostic Test: Point-of-care hepatitis C antibody test; Diagnostic Test: Point-of-care hepatitis C RNA test; Diagnostic Test: Point-of-care hepatitis B surface antibody test; Diagnostic Test: Point-of-care hepatitis B surface antigen test; Diagnostic Test: Point-of-care HIV antibody test; Behavioral: Interview-style survey

INTERVENTIONS:
Diagnostic Test: Point-of-care hepatitis C antibody test — Qualitative point-of-care test for hepatitis C antibodies (saliva sample)
  Other Names: OraQuick HCV Rapid Antibody Test
Diagnostic Test: Point-of-care hepatitis C RNA test — Hepatitis C Viral Load point-of-care test (fingerstick wholeblood sample)
  Other Names: Xpert HCV VL Fingerstick
Diagnostic Test: Point-of-care hepatitis B surface antibody test — Qualitative hepatitis B surface antibody point-of-care test (fingerstick wholeblood sample)
  Other Names: QuickProfile HBsAb Fingerstick test
Diagnostic Test: Point-of-care hepatitis B surface antigen test — Qualitative hepatitis B surface antigen point-of-care test (fingerstick wholeblood sample)
  Other Names: Alere Determine 2 HBsAg Fingerstick Test
Diagnostic Test: Point-of-care HIV antibody test — Qualitative HIV antibody point-of-care test (saliva sample)
  Other Names: OraQuick Rapid ADVANCE HIV 1/2 Antibody Test
Behavioral: Interview-style survey — Interview-style survey regarding demographics, risk behaviours, BBV testing and treatment history, and point-of-care testing acceptability

SUMMARY:
The Australian Hepatitis and risk survey in prisons (AusHep) is a national prison-based blood-borne virus (BBV) surveillance study. This biobehavioural survey involves point-of-care testing for hepatitis C (HCV) antibodies and RNA (if antibody positive), hepatitis B surface antigens, hepatitis B surface antibodies, and HIV surface antibodies, and an interview-style survey on prior testing and treatment history and engagement in risk behaviours. The study will recruit approximately 2400 prisoner participants from 25 representative prisons across Australia, annually.

ELIGIBILITY:
Inclusion Criteria:

* Any remandee or sentenced prisoner who has provided informed consent is eligible to participate in the study.

Exclusion Criteria:

* Individuals who are unable or unwilling to provide consent or abide by the requirements of the study, as assessed by the trained nurses. Some individuals may be considered unable to provide consent or abide by the requirements of the study if they are:

  * Too mentally unwell to provide consent
  * Profoundly intellectually impaired
  * Unable to speak English and comprehend the survey.

Those excluded from participating in the study will be referred to the local prison clinic service for standard of care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the selected correctional centre(s) in each jurisdiction. All prisoners, including remandees and sentenced prisoners at the selected site(s) will be randomly selected to participate.
Sampling Method: Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2022-04-27 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
The prevalence of HCV in Australian prisons | 1 Year
  This is estiamted by perfroming the HCV antibody test and HCV RNA viral load test on a representative prison population.
The prevalance of HBV in Australian prisons | 1 year
  This is estimated by performing the HBV surface antigen test on a respresentative prison population
The prevalance of HIV in Australian prisons | 1 year
  This is estimated by performing the HIV antibody test on a respresentative prison population.

SECONDARY OUTCOMES:
The proportion of individuals who are engaged in each step of HBV and HCV care cascades | 1 Year
  This is estimated by conducting the bio-behavioural survey.
The prevalence of risk behaviours and harm reduction access | 1 Year
  The risk behavrious and harm reduction measures include injecting and non-injecting drug use, high risk injecting practices, sexual risk behaviours, tattooing; and bleach or opioid substitution therapy (OST) uptake. This is estimated by conducting the bio-behavioural survey.
The factors associated with HCV and HBV infection investigated by the bio-behavioural survey. | 1 Year
The factors associated with engaging in each step of HCV and HBV care cascades and HBV vaccination investigated by the bio-behavioural survey. | 1 Year

CONTACTS AND LOCATIONS:
Locations (24):
- Australia (24):
  - Alexander Maconochie Centre, Hume, Australian Capital Territory
  - Bathurst Correctional Complex, Bathurst, New South Wales
  - John Morony Correctional Complex, Berkshire Park, New South Wales
  - Cessnock Correctional Centre, Cessnock, New South Wales
  - Mid North Coast Correctional Centre, Kempsey, New South Wales
  - South Coast Correctional Centre, Nowra, New South Wales
  - Silverwater Women's Correctional Centre, Silverwater, New South Wales
  - Wellington Correctional Centre, Wuuluman, New South Wales
  - Alice Springs Correctional Centre, Alice Springs, Northern Territory
  - Darwin Correctional Centre, Howard Springs, Northern Territory
  - Borallon Training and Correctional Centre, Ironbark, Queensland
  - Brisbane Women's Correctional Centre, Ironbark, Queensland
  - Wolston Correctional Centre, Ironbark, Queensland
  - Townsville Correctional Centre, Townsville, Queensland
  - Mobilong Prison, Murray Bridge, South Australia
  - Adelaide Women's Prison, Northfield, South Australia
  - Yatala Labour Prison, Northfield, South Australia
  - Mary Hutchinson Women's Prison, Risdon Vale, Tasmania
  - Risdon Maximum Prison, Risdon Vale, Tasmania
  - Ron Barwick Minimum Security Prison, Risdon Vale, Tasmania
  - Bunbury Regional Prison, Bunbury, Western Australia
  - Casuarina Prison, Casuarina, Western Australia
  - Roebourne Regional Prison, Roebourne, Western Australia
  - Bandyup Women's Prison, West Swan, Western Australia

IPD SHARING:
Plan to Share IPD: No